CLINICAL TRIAL: NCT00795457
Title: A Bi-Institutional Pilot Study to Evaluate the Effects of Vaccinations With HLA-A2-Restricted Glioma Antigen-Peptides in Combination With Poly-ICLC for Adults With WHO Grade II Low-Grade Gliomas
Brief Title: Effects of Vaccinations With HLA-A2-Restricted Glioma Antigen-Peptides in Combination With Poly-ICLC for Adults With High-Risk WHO Grade II Astrocytomas and Oligo-Astrocytomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ian F. Pollack, M.D. (Other)
Collaborators: Oncovir, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ian F. Pollack, M.D., Chief, Pediatric Neurosurgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-057; R21CA133859-01A1 (NIH)
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Astrocytoma; Oligo-Astrocytoma; Glioma
Keywords: vaccine; WHO Grade II Astrocytoma; WHO Grade II Oligo-Astrocytoma
MeSH Terms: conditions — Astrocytoma; Glioma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients must have undergone surgery or biopsy alone ≤16 weeks prior to study entry (no postoperative radiation or chemotherapy).
  Interventions: Biological: GAA/TT-peptide vaccine and poly-ICLC
- 2 (Experimental): Patients received surgery or biopsy and radiation therapy (RT) (including fractionated external beam radiation therapy and/or stereotactic radiosurgery), which was completed ≥6 months prior to enrollment, and have a baseline MRI scan (within 4 weeks of the first vaccine) that shows stable disease or regression.
  Interventions: Biological: GAA/TT-peptide vaccine and poly-ICLC

INTERVENTIONS:
Biological: GAA/TT-peptide vaccine and poly-ICLC — Participants will be treated with subcutaneous injections of GAA/TT-vaccines on Weeks 0, 3, 6, 9, 12, 15, 18 and 21. I.m. poly-ICLC will be administered (20 mg/kg i.m.) on the day of, and on day 4 after each vaccine (e.g. if the vaccine is administered on Thursday, poly-ICLC will be administered on the day of vaccine and the following Monday). Each vaccine will be administered within 2 hours before or after the i.m. poly-ICLC administration.
  Arms: 1
Biological: GAA/TT-peptide vaccine and poly-ICLC — Participants will be treated with subcutaneous injections of GAA/TT-vaccines on Weeks 0, 3, 6, 9, 12, 15, 18 and 21. I.m. poly-ICLC will be administered (20 mg/kg i.m.) on the day of, and on day 4 after each vaccine (e.g. if the vaccine is administered on Thursday, poly-ICLC will be administered on the day of vaccine and the following Monday). Each vaccine will be administered within 2 hours before or after the i.m. poly-ICLC administration.
  Arms: 2

SUMMARY:
This is a pilot vaccine study in adults with either WHO grade II astrocytoma, oligoastrocytoma or oligodendroglioma. The purpose of this study is test the safety and efficacy of an experimental tumor vaccine made from peptides and Montanide ISA-51 in combination with the study drug Poly-ICLC.

Poly-ICLC, manufactured by Oncovir, Inc., has already been received and generally well tolerated by subjects in earlier studies and has been shown to decrease the size of brain tumors in some cases.

The immunological and safety data will be used to decide whether a larger study of clinical efficacy is warranted in each of two patient cohorts.

DETAILED DESCRIPTION:
All patients on the study will be followed for a minimum of 2 years, so that the actual 2-year overall survival (OS) and progression-free survival (PFS) rates can be determined in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have documented pathological diagnosis of a WHO grade II astrocytoma or oligoastrocytoma or oligodendroglioma (see also the 4th bullet for oligodendroglioma).
* HLA-A2 positive based on flow cytometry.
* There will be 2 cohorts of patients based on whether patients have received prior RT. Cohort 1: patients must have undergone surgery or biopsy alone ≤16 weeks prior to study entry (no postoperative radiation or chemotherapy). Cohort 2: Patients received surgery or biopsy and radiation therapy (RT) (including fractionated external beam radiation therapy and/or stereotactic radiosurgery), which was completed ≥6 months prior to enrollment, and have a baseline MRI scan (within 4 weeks of the first vaccine) that shows stable disease or regression.
* For oligodendroglioma, at least one of the following three conditions has to be met: 1) age ≥ 40 with any extent resection; 2) age 18-39 with incomplete resection (post-op MRI showing > 1cm residual disease, based on the maximum dimension of residual T2 or FLAIR abnormality from the edge of the surgical cavity either laterally, antero-posteriorly, or supero-inferiorly) or 3) age 18-39 with neurosurgeon-defined GTR but the tumor size is ≥ 4 cm (the maximum preoperative tumor diameter, based on the axial and/or coronal T2 or FLAIR MR images). Participants must be ≥ 18 years old because the safety of each therapeutic component has not been established in children.
* All participants must sign an informed consent document indicating that they are aware of the investigational nature of this study.
* Participants must have a Karnofsky performance status of > 60 (Appendix I).
* Documented negative serum beta HCG for female participants of child-bearing age. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the peptide based vaccine and poly-ICLC, breastfeeding should be discontinued if the mother is treated in this study.
* Participants must be free of systemic infection
* Participants with adequate organ function as measured by white blood count ≥ 2500/mm3; lymphocytes ≥ 800/mm3; platelets ≥ 100,000/mm3, hemoglobin ≥ 10.0 g/dL, AST, ALT, GGT, LDH, alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin greater than or equal to 2.0 mg/dL, and serum creatinine within 1.5 X upper limit of normal limit. Coagulation tests PT and PTT have to be within normal limits.

Exclusion Criteria:

* Presence of cranial or spinal leptomeningeal metastatic disease.
* Prior chemotherapy or anti-glioma therapy of any type other than radiation therapy (see 3.1.3)
* Concurrent treatment or medications including:

  * Radiation therapy
  * Chemotherapy
  * Interferon
  * Allergy desensitization injections
  * Growth factors
  * Interleukins
  * Any investigational therapeutic medication
* Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. Mild arthritis requiring NSAID medications will not be exclusionary.
* Use of immunosuppressives within 4 weeks prior to study entry or anticipated use of immunosuppressive agents. Dexamethasone, or other corticosteroid medications, if used perioperative period and/or during radiotherapy, must be tapered and discontinued at least 4 weeks before administration of the first vaccine. Topical corticosteroids and Inhaled steroids are acceptable.
* Participants who have another cancer diagnosis, except that the following diagnoses will be allowed:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
  * any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 5 years
* Participants with known addiction to alcohol or any drugs.
* Because patients with immune deficiency are not expected to respond to this therapy, HIV positive patients are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Induction of GAA-specific T-cell response | 2 year
The incidence and severity of adverse events associated with the vaccine regime will be assessed, with an early stopping rule based on the frequency of Regimen Limiting Toxicity (RLT). | 1 year

SECONDARY OUTCOMES:
Clinical Response: Radiological response will be determined using the standard WHO response criteria. Based on serial magnetic resonance imaging (MRI) scans 2-year progression-free survival (PFS) will be evaluated in an exploratory manner. | 3 years
Biopsy/resection will be encouraged for patients who develop progression. Whenever post-vaccine tumor tissues are available, they will be analyzed for GAA expression status and infiltration of GAA-specific T-cells. | 3 years
Influence of RT on induction of GAA-specific immune response: we will compare the rate and magnitude of GAA-specific immune responses in Cohorts 1 and Cohort 2 using IFN-gamma-enzyme-linked immuno-spot (ELISPOT), and tetramer assays. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lieberman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania